CLINICAL TRIAL: NCT04762823
Title: Multiple Sessions of Transcranial Direct Current Stimulation in People With Parkinson's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI (Post-Doc Craig Workman) left the university.
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202007551
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Parkinson Disease; Healthy Adult
Keywords: transcranial direct current stimulation; cerebellum; gait; balance; cognition; fatigue
MeSH Terms: conditions — Parkinson Disease; Fatigue

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Subjects will be blind to the different stimulation intensities (sham, 4 mA) and the test administrators will also be blind to the subject's assigned stimulation condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- PD-ctDCS (Experimental): People with Parkinson's disease will have both electrodes placed 1-2 cm below and 3 cm to either side of the inion, with the anode assigned to the most PD-affected side and the cathode assigned to the less PD-affected side. Stimulation is ramped up to 4 mA over the first 30 seconds and stays at 4 mA for the remainder of the stimulation time.
  Interventions: Device: Cerebellar transcranial direct current stimulation at 4 mA
- PD-sham (Sham Comparator): People with Parkinson's disease will have both electrodes placed 1-2 cm below and 3 cm to either side of the inion, with the anode assigned to the most PD-affected side and the cathode assigned to the less PD-affected side. Stimulation is turned on (4 mA) for 30 seconds at the beginning and the end of the trial, but it turned to 0 mA in the intervening time.
  Interventions: Device: Sham cerebellar transcranial direct current stimulation
- NH-ctDCS (Active Comparator): Neurologically healthy older adults will have both electrodes placed 1-2 cm below and 3 cm to either side of the inion, with the anode assigned to the most PD-affected side and the cathode assigned to the non-dominant side. Stimulation is ramped up to 4 mA over the first 30 seconds and stays at 4 mA for the remainder of the stimulation time.
  Interventions: Device: Cerebellar transcranial direct current stimulation at 4 mA
- NH-sham (Sham Comparator): Neurologically healthy older adults will have both electrodes placed 1-2 cm below and 3 cm to either side of the inion, with the anode assigned to the most PD-affected side and the cathode assigned to the non-dominant side. Stimulation is turned on (4 mA) for 30 seconds at the beginning and the end of the trial, but it turned to 0 mA in the intervening time.
  Interventions: Device: Sham cerebellar transcranial direct current stimulation

INTERVENTIONS:
Device: Cerebellar transcranial direct current stimulation at 4 mA — Uses weak electrical current (4 mA intensity) to either increase or decrease brain excitability and improve functional or cognitive outcomes.
  Other Names: ctDCS
  Arms: NH-ctDCS; PD-ctDCS
Device: Sham cerebellar transcranial direct current stimulation — Uses weak electrical current (4 mA intensity) at the beginning and the end of a given stimulation period to control for potential placebo effects or participant expectation bias.
  Other Names: Sham
  Arms: NH-sham; PD-sham

SUMMARY:
Parkinson's disease (PD) affects approximately 1 million people in the US, with annual health care costs approaching $11 billion. PD results from a loss of dopamine-producing cells in the brain. This decrease in dopamine is associated with shaking, stiffness, slowness, balance/walking problems, thinking, and fatigue which severely impair activities of daily living. Current medical and surgical treatments for PD are either only mildly effective, expensive, or associated with a variety of side-effects. Therefore, the development of practical and effective therapies would have significant benefits.

Transcranial direct current stimulation (tDCS) can influence how the brain works. A review of studies concluded that, overall, tDCS improves walking and balance in people with PD (PwPD). However, these studies had mixed results. For example, most have stimulated the frontal brain areas and all have used intensities of 2 mA (milliamperes; a measure of electrical current strength) or less. However, given the vital role of the cerebellum in walking and balance, and in PD impairments, the cerebellum may represent a more effective brain target. A recent review of studies also recommended performing investigations of higher intensity tDCS (greater than 2 mA), to potentially increase stimulation efficacy. No study has investigated the effects of multiple sessions of cerebellar tDCS on gait and balance in PwPD and none have used tDCS intensities greater than 2 mA. Therefore, there is a critical need to determine if repeated sessions of cerebellar tDCS might improve walking and balance in the short- and long-term.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, people with PD must meet the following criteria:

1. Adult (50-90 yrs) with a positive diagnosis of Parkinson's disease from a movement disorder specialist
2. On an unchanged regimen of dopaminergic medication for at least the last 3 months
3. Able to independently walk for 6 min
4. Without other severe chronic psychiatric or medical conditions
5. Not taking any psychoactive medications

To be eligible to participate in this study, the NH subjects must meet the following criteria:

1. Adult (50-90 yrs)
2. Able to independently walk for 6 min
3. Without any severe chronic psychiatric or medical conditions
4. Not taking any psychoactive medications

Exclusion Criteria:

An individual from either group who meets any of the following criteria will be excluded from participation in this study:

1. Pregnant
2. Known holes or fissures in the skull
3. Metallic objects or implanted devices in the skull/head (e.g., metal plate, deep brain stimulator)
4. Current or previous injuries or surgeries that cause unusual gait
5. A score less than 24 or 17 on the Montreal Cognitive Assessment (MoCA) or telephone-MoCA, respectively

Additional exclusion for PwPD:

1. Experience freezing of gait
2. A diagnosis of dementia or other neurodegenerative diseases

Additional exclusion for NH subjects:

1. A diagnosis of dementia or any neurodegenerative diseases

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-15 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society version of the Unified Parkinson's Disease Rating Scale (MDS-UPRDS) | Through study completion, up to 12 months
  The scale includes four parts that assess activities of daily living (Parts I and II), a motor exam (Part III), and medication-related motor complications (Part IV). For all parts, a higher number indicates more disability.
Fatigue Severity Scale (FSS) | Through study completion, up to 12 months
  A nine-item questionnaire asking subjects to rate the severity of their perceived fatigue on a 1-7 point Likert scale (a higher number means more subjective fatigue).
Multidimensional Fatigue Inventory (MFI) | Through study completion, up to 12 months
  A 20-item scale evaluating five dimensions of fatigue rated on a 1-5 point Likert scale (positively phrase items reverse scored; a higher number means more fatigue).
30-meter walk test, single-task (30mWT-ST; 2 trials) | Through study completion, up to 12 months
  Subjects walk at their usual/comfortable speed; walking characteristics and the time taken to complete the task are the primary outcomes (more time = worse performance)
30-meter walk test, dual-task (30mWT-DT; 2 trials) | Through study completion, up to 12 months
  Same as 30mWT-ST, except the subjects perform a secondary/cognitive task during the walking. The secondary task will involve serially subtracting 7 from a randomly selected starting number (100, 125, 150, 200; won't repeat a starting number within a given session). Changes in task performance between single- and dual-task conditions represent dual-task interference.
6-minute walk test (6MWT; 1 trial) | Through study completion, up to 12 months
  Subjects walk back and forth between two markers spaced 30 m apart at the usual speed. The total distance walked is the primary outcome (longer distance walked is an analog for less fatigue).
9-hole peg test (9-HPT; two trials with each hand) | Through study completion, up to 12 months
  The subjects are instructed to pick up the pegs from a shallow cup one at a time, place them in the holes, and then immediately take the pegs back out of the holes one at a time. Time to put the pegs in and take them out again is recorded (more time = worse performance).
Reaction time test (simple and choice; 1 trial each) | Through study completion, up to 12 months
  Simple: A white box is displayed on a computer screen. When a black X appears in the white box, the subjects need to press the computer space bar as quickly as possible. Several trials with random inter-stimulus-intervals are presented. Choice: Four white boxes are displayed on the screen. When a black X appears in one of the boxes, the subjects need to press the appropriate key (z = left-most box, x = second from left, comma (,) = third from left, and period (.) = right-most) as quickly as possible. The average reaction time is recorded (more time = worse performance).
Flanker Inhibitory Control and Attention Test (1 trial) | Through study completion, up to 12 months
  On each trial, a central directional target (arrow) is flanked by similar stimuli on the left and right (five total arrows). The task is to indicate the direction of the central stimulus (i.e., the third arrow). On congruent trials, the flanker arrows face the same direction as the target. On incongruent trials, they face the opposite direction. Time to react to the different conditions is recorded (more time = worse performance).
Trail Making Test A and B (TMT A/B; 1 trial each) | Through study completion, up to 12 months
  Both parts consist of 25 circles (Part A: numbered 1 - 15; Part B: numbers and letters 1- 13 and A - L). The subject draws lines connecting the numbers in ascending order (Part A: 1-2-3-4-5 etc.) and then in alternating-ascending order (Part B; e.g., 1-A-2-B-3-C, etc.) as quickly and as accurately as possible without lifting the pen/pencil off the paper. Time to complete the "trail" is recorded (more time = worse performance).
Berg Balance Scale (BBS) | Through study completion, up to 12 months
  14-item scale rated on a 0 - 4 Likert scale that assesses balance performance in several dynamic and static conditions (lower score = worse balance).
Static Posturography. | Through study completion, up to 12 months
  1) stand on a firm surface (directly on a force platform) for 1 minute with eyes open (balance characteristics [95% confidence interval of the total 2D area explored, the center of pressure movement velocity in forward/backward and left/right directions] are the primary outcomes), 2) stand on a foam surface (6 cm foam pad placed on top of force platform) for 1 minute with eyes open (the same balance characteristics as above are the primary outcomes).

SECONDARY OUTCOMES:
Brain activity PET Imaging with [18F]Fluorodeoxyglucose (FDG) | Through study completion, up to 12 months
  Assesses resting-state brain activity by determining brain glucose usage. Involves the injection of a radioactive glucose analog that can be imaged with the PET scanner.

CONTACTS AND LOCATIONS:
Overall Officials: Craig D Workman, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No